CLINICAL TRIAL: NCT05231798
Title: Cholinergic Integrity in Down Syndrome in Association With Aging, Alzheimer's Disease Pathology, and Cognition
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Vanderbilt Kennedy Center (Other)
Responsible Party: Principal Investigator, Alexander Christian Conley, PhD, Principal Investigator, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 210933
Record Dates: First submitted 2022-01-17; First posted 2022-02-09 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-03

CONDITIONS: Down Syndrome; Down Syndrome, Partial Trisomy 21; Alzheimer Disease
MeSH Terms: conditions — Down Syndrome; Alzheimer Disease | interventions — fluoroethoxy-benzovesamicol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Down Syndrome (Experimental): Adults between 18-55 with Down Syndrome.
  Interventions: Drug: [18F]-FEOBV Radiotracer

INTERVENTIONS:
Drug: [18F]-FEOBV Radiotracer — Participants will be administered an [18F]-fluoroethoxybenzovesamicol (FEOBV) radiotracer for diagnostic imaging purposes (PET scan).
  Other Names: [18F]-fluoroethoxybenzovesamicol

SUMMARY:
Progressive age-related cognitive deficits occurring in both AD and DS have been connected to the degeneration of several neuronal populations, but mechanisms are not fully elucidated. The most consistent neuronal losses throughout the progression of AD are seen in cholinergic neurons where these losses negatively affect cognition, particularly in attention, learning, and memory formation. Evidence of reduced cholinergic integrity in DS is largely limited to animal models and post-mortem human data. The investigators propose to use molecular, functional, and structural biomarkers to assess the cholinergic integrity in adults with DS. The investigators anticipate using the data gathered in this pilot study to inform future study designs to determine AD risk stratification in DS by identifying individuals who show an accelerated decline in cholinergic integrity that correlates with cognitive and neurobehavioral changes. Also, our cholinergic biomarkers may identify whether individuals with DS are likely to respond to pro-cholinergic interventions, including the novel cholinergic modulators that are being developed to enhance cholinergic-sensitive cognitive functioning. The investigators anticipate using the data gathered here to inform future treatment studies in TRC-DS and beyond where novel cholinergic treatments may offer opportunities for early intervention in DS and be complementary to disease-modifying approaches such as anti-amyloid treatments.

DETAILED DESCRIPTION:
Down syndrome (DS) or Trisomy 21, is the most common genetic cause of intellectual disability. Among its consequences, by the age of 30, people with DS invariably develop amyloid plaques and neurofibrillary tangles such that up to 75% of people with DS will develop Alzheimer's disease (AD). AD in DS is thought to be linked to the presence of three copies of the amyloid precursor protein (APP) gene, which resides on chromosome 21. This gene leads to higher levels of amyloid-β (Aβ) plaques. Preliminary data show that adults with DS exhibit significant changes in AD-related biomarkers between the ages of 35-55. It is also within this age range that AD-related cognitive decline and dementia typically manifest in DS. AD is the primary cause of death in adults with DS over the age of 35. Although it is currently suggested that the onset of dementia in DS is in part due to triplication of the amyloid precursor protein (APP) gene, other neurodegenerative features of sporadic AD may occur in DS and these can aggravate the onset of cognitive decline and dementia. Progressive cognitive deficits occurring in sporadic AD are associated with the degeneration of several neuronal populations. Throughout the progression of AD, the most consistent losses are seen in cholinergic neurons. While the loss of the cholinergic integrity has been established as a critical biological process in sporadic AD, the cholinergic system has not been evaluated in adults with DS to examine if age-related cholinergic decline can be detected in DS and whether it is associated with the progression of AD pathologies and cognitive decline as seen in sporadic AD.

The investigators propose to conduct a pilot study that aims to assess the integrity of the cholinergic neurotransmission system using in-vivo structural, functional, and molecular imaging biomarkers.

The examination of the cholinergic system in DS and its relationship to aging and known AD pathologies and cognitive decline would help validate whether the cholinergic decline is an early marker of dementia risk in DS and proceeds or follows changes in standard AD imaging and fluid biomarkers, thus helping establish how similar AD in DS is to that of sporadic AD. The investigators anticipate using the data gathered here to inform future treatment studies where novel cholinergic treatments may offer opportunities for early intervention in DS and be complementary to disease-modifying approaches such as anti-amyloid treatments.

Objective: To examine the molecular, functional, and structural biomarkers of cholinergic integrity in Down syndrome (DS) in association with age, Alzheimer's disease (AD) pathology, and cognitive/neurobehavioral performance.

Specific Aim: The Center for Cognitive Medicine is a site for the Trial-Ready Cohort-Down Syndrome (TRC-DS) study, to enable a systematic biomarker characterization of middle-aged and older individuals with DS by using neuroimaging, cognitive, and clinical measures, in preparation for an AD-like prevention trial likely using anti-amyloid agents. The investigators will leverage this cohort's well-characterized DS participants to initiate a new pathway for investigating our novel cholinergic biomarker in 10 TRC-DS participants (age:35-55) and enroll 110 additional adults with DS (age:18-55) outside of the TRC-DS study.

The investigators will use molecular, functional, and structural biomarkers to measure the cholinergic integrity of adults with DS. These methods will include resting and task-related electroencephalogram (EEG), basal forebrain volumetric measures on structural magnetic resonance imaging (MRI), and positron emission tomography (PET) with a vesicular cholinergic radiotracer known as fluoroethoxybenzovesamicol ([18F]FEOBV).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Down syndrome (DS), including mosaic DS or partial trisomy 21.
2. Provision of signed and dated informed consent form and if needed, assent with signed consent by a legally authorized representative (LAR).
3. Stated willingness to comply with all study procedures and availability for the duration of the study
4. Male or female, aged 18-55 inclusive.
5. In good general health as evidenced by medical history with no diagnosis of dementia.
6. Permitted CNS-active medications, stable in dose for at least 4 weeks or longer. If new medications have been started, the medical monitoring team will review on case-by-case basis to recommend timing of baseline cognitive testing
7. Adequate visual and auditory acuity to allow neuropsychological testing
8. For females who are not surgically sterile or post-menopausal by two years: negative pregnancy test 24 hours prior to PET scan.
9. Mental Age of 4 years or greater (based upon the Kaufman Brief Intelligence Test, 2nd Edition)
10. English must be first/native language
11. Reliable Study Partner (may be caregiver, sibling, parent) who can provide information about the subject's clinical symptoms and history

Exclusion Criteria:

1. Any significant disease or unstable medical condition that could affect neuropsychological testing (i.e., unstable cardiac problems, chronic renal failure, chronic hepatic disease, severe pulmonary disease)
2. Participants in whom magnetic resonance imaging (MRI) is contraindicated including, but not limited to, those with a pacemaker, presence of metallic fragments near the eyes or spinal cord, or cochlear implant (Dental fillings do not present a risk for MRI)
3. Participants unable to complete MRI and PET procedures
4. IQ less than 40 (as assessed by Kaufman Brief Intelligence Test, Second Edition (KBIT-2).
5. Pregnancy, breast-feeding
6. History within the last 5 years of a primary or recurrent malignant disease with the exception of non-melanoma skin cancers, resected cutaneous squamous cell carcinoma in situ, basal cell carcinoma, cervical carcinoma in situ, or in situ prostate cancer with normal prostate-specific antigen post-treatment
7. Clinically significant abnormalities in B12 or TFTs that might interfere with the study. A low B12 is exclusionary unless follow-up labs (homocysteine (HC) and methylmalonic acid (MMA)) indicate that it is not physiologically significant. A high TSH is exclusionary unless follow-up T3/T4 levels indicate that it is not physiologically significant.
8. Clinically significant abnormalities in screening laboratories
9. For participants undergoing CSF collection: a current blood clotting or bleeding disorder, or significantly abnormal PT or PTT at screening or if on anti-coagulation (e.g warfarin)
10. Participants whom the Site PI deems to be otherwise ineligible
11. Clinical diagnosis of dementia
12. Concurrent participation in a clinical trial for an investigational product or concurrent participation in a longitudinal study with overlapping outcome measures/procedures is prohibited

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
[18F]-FEOBV radiotracer standardized uptake value ratio correlation with the Basal Forebrain Cholinergic System Volume. | Analysis will be completed at study completion in approximately 3 years.
  The association of [18F]-FEOBV radiotracer standardized uptake value ratio with the the gray matter volume of the cholinergic basal forebrain in adults with Down syndrome.

SECONDARY OUTCOMES:
EEG resting state power correlation with [18F]-FEOBV radiotracer standardized uptake value ratio | Analysis will be completed at study completion in approximately 3 years.
  The association of EEG resting state power with [18F]-FEOBV radiotracer standardized uptake value ratio in adults with Down syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander C Conley, Ph.D., Principal Investigator — Vanderbilt University Medical Center; Paul A Newhouse, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center Clinical Research Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be available upon request.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will become available after the study completion, anticipated to be 08/19/2024
Access Criteria: Access will be granted to qualified individuals upon request.